CLINICAL TRIAL: NCT00524225
Title: Phase II Clinical Efficacy Trial of Recombinant Interleukin-11 (rhIL-11, Neumega) in Subjects With Type 1 Von Willebrand Disease Undergoing Surgery
Brief Title: IL-11 in Adults With Von Willebrand Disease Undergoing Surgery
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Recruitment slow as single center conducting in rare disease
Sponsor: Margaret Ragni (Other)
Collaborators: University of North Carolina (Other); Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Sponsor-Investigator, Margaret Ragni, Professor, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: PRO07030210
Record Dates: First submitted 2007-08-31; First posted 2007-09-03 (Estimated); Results first posted 2014-11-07 (Estimated); Last update posted 2019-06-11 (Actual); Status verified 2019-06

CONDITIONS: Von Willebrand Disease
Keywords: IL-11; von Willebrand disease; von Willebrand factor; VWFmRNA; surgery
MeSH Terms: conditions — von Willebrand Diseases | interventions — oprelvekin; Interleukin-11

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Neumega (Interleukin 11, IL-11) (Experimental): Neumega (Oprelvekin, Interleukin 11, IL-11) 25 mcg/kg subcutaneously, given for 4 days preoperatively, and on day 5 preoperatively, and for up to 2 days postoperatively
  Interventions: Drug: Neumega (Oprelvekin, Interleukin 11, IL-11)

INTERVENTIONS:
Drug: Neumega (Oprelvekin, Interleukin 11, IL-11) — 25 micrograms/kg by subcutaneous injection once daily for four days, followed by once daily on days 1-3 before and after elective surgery or dental procedure

SUMMARY:
The purpose of this study is to determine the efficacy and safety of rhIL-11 when given subcutaneously in adults with type 1 von Willebrand disease undergoing elective surgery or major dental procedure. Efficacy will be measured by estimated blood loss, and frequency and severity of bleeding and transfusion requirement during and after surgery. Safety will be measured by the frequency of adverse events, including fever, headache, fatigue, myalgias, arthralgias, fluid retention, or edema.

DETAILED DESCRIPTION:
This study is a prospective, single-center Phase II trial of Neumega (rhIL-11) in adults with type 1 VWD undergoing elective surgery or major dental procedure. It is anticipated that 10 subjects who meet eligibility criteria will enroll and complete the study. The specific objectives are to determine the efficacy and safety or rhIL-11 during and after elective surgery, and to determine the mechanism of the hemostatic response of rhIL-11.

ELIGIBILITY:
Inclusion Criteria:

* Males and females 18 years of age and older
* Confirmed type 1 VWD, as defined by low VWF:RCoF or low VWF:Ag and qualitatively normal VWF multimers
* A past bleeding history
* Responsive to DDAVP
* Scheduled elective major surgery or major dental surgery at MUH or PUH
* Willingness to have blood drawn

Exclusion Criteria:

* Presence of other bleeding disorders, acquired Von Willebrand disease, primary thrombocytopenia
* Use of immunomodulatory or experimental drugs, or diuretics
* Pregnant or lactating women or those unwilling to use contraception during study
* Previous cardiac disease, congestive failure, arrhythmia (e.g. atrial fibrillation, atrial flutter), hypertension, MI, stroke, or thrombosis
* Past allergic reaction to Neumega or DDAVP
* Surgery within the past 8 weeks
* Inability to comply with study protocol requirements
* Concomitant use of antiplatelet drugs, anticoagulants, dextran, aspirin or NSAIDs
* Treatment with DDAVP, cryoprecipitate, whole blood, plasma and plasma derivatives containing substantial quantities of FVIII and/or VWF within five days of study
* Past allergic reaction to Neumega or DDAVP
* Surgery within the past 8 weeks
* Inability to comply with study protocol requirements
* Concomitant use of antiplatelet drugs, anticoagulants, dextran, aspirin or NSAIDs
* Treatment with DDAVP, cryoprecipitate, whole blood, plasma and plasma derivatives containing substantial quantities of FVIII and/or VWF within five days of study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2008-02; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Margaret V Ragni, MD, MPH, Principal Investigator — University of Pittsburgh Medical Center
Locations (1):
- Hemophilia Center of Western PA, Pittsburgh, Pennsylvania, United States

REFERENCES:
- [Background] Jankowitz RC, Nichols TC, Ragni MV. Recombinant IL-11 (Neumega, rhIL-11) increases plasma Von Willebrand Factor in Type 1 Von Willebrand Disease. Blood 108: 1003, 2006 (abstract).
- [Background] Ragni MV, Jankowitz RC, Chapman HL, Merricks EP, Kloos MT, Dillow AM, Nichols TC. A phase II prospective open-label escalating dose trial of recombinant interleukin-11 in mild von Willebrand disease. Haemophilia. 2008 Sep;14(5):968-77. doi: 10.1111/j.1365-2516.2008.01827.x. Epub 2008 Aug 1. PMID 18680527

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Neumega (Interleukin 11, IL-11)
Started | 3
Completed | 3
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Neumega (Interleukin 11, IL-11)
Number analyzed (Participants) | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 3
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 0

OUTCOME MEASURES:

1. Primary Outcome: Volume of Surgical Blood Loss
Description: Hemostatic efficacy was measured by estimated blood loss (cc) during the surgical procedure.
Time Frame: 4 weeks
Measure: Number; unit: cc
Arm/Group | Neumega (Interleukin 11, IL-11)
Number analyzed (Participants) | 3
cc | NA — Volume of surgical blood loss was negligible for all participants.

2. Primary Outcome: Volume of Blood Transfusion
Description: The volume of blood transfusion required (units of blood) after the surgical procedure.
Time Frame: 4 weeks
Measure: Number; unit: units of blood
Arm/Group | Neumega (Interleukin 11, IL-11)
Number analyzed (Participants) | 3
units of blood | NA — No participant had a transfusion.

3. Secondary Outcome: No. of Subjects With Detectable VWFmRNA (Von Willebrand Factor Messenger RNA).
Description: The number of subjects with detectable VWFmRNA.
Time Frame: 4 weeks per subject
Population: Even though three subjects were enrolled, none were assessed for VWFmRNA because the study stopped due to poor enrollment related to insurers requiring surgeries outside of UPMC.
Arm/Group | Neumega (Interleukin 11, IL-11)
Number analyzed (Participants) | 0

4. Secondary Outcome: Number of Subjects Who Experienced Adverse Events
Description: mild headache, nausea
Time Frame: The time frame is within 4 weeks of surgery.
Measure: Number; unit: participants
Arm/Group | Neumega (Interleukin 11, IL-11)
Number analyzed (Participants) | 3
participants
  Mild headache | 1
  nausea | 1

ADVERSE EVENTS:
Arm/Group | Neumega (Interleukin 11, IL-11)
Serious Adverse Events (participants affected / at risk) | 0/3
Other Adverse Events (participants affected / at risk) | 2/3
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Neumega (Interleukin 11, IL-11) (N=3)
headache (Nervous system disorders) | 1 (1) — mild headache
nausea (Gastrointestinal disorders) | 1 (1) — mild nausea

LIMITATIONS AND CAVEATS:
There were too few subjects for reporting in a manuscript.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes